CLINICAL TRIAL: NCT02290938
Title: Motivational Interviewing and Culture for Urban Native American Youth (MICUNAY)
Acronym: MICUNAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute on Drug Abuse (NIDA) (NIH); University of California, Los Angeles (Other); Sacred Path Indigenous Wellness Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AA022066 (NIH); 1R01AA022066 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-11-14 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use; Marijuana Use
Keywords: adolescents; Native American; alcohol use; drug use; cultural; traditional activities; cultural identification
MeSH Terms: conditions — Alcohol Drinking; Marijuana Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community Wellness Gatherings (Active Comparator): All youth will attend a CWG, which is a monthly gathering focused on making healthy choices and learning about Native American culture
  Interventions: Other: Community Wellness Gathering
- Community Wellness Gathering + MICUNAY (Experimental): MICUNAY is a three session workshop focused on discussions about how to make healthy choices using motivational interviewing, and providing a cultural activity.
  Interventions: Behavioral: MICUNAY

INTERVENTIONS:
Behavioral: MICUNAY — MICUNAY is a three session workshop focused on discussions about how to make healthy choices using motivational interviewing, and providing a cultural activity.
  Arms: Community Wellness Gathering + MICUNAY
Other: Community Wellness Gathering — a monthly gathering focused on making healthy choices and learning about Native American culture
  Arms: Community Wellness Gatherings

SUMMARY:
The investigators plan to develop and test a new alcohol and other drug (AOD) intervention for urban AI/AN youth, "Motivational Interviewing and Culture for Urban Native American Youth (MICUNAY)." This intervention integrates tradition-based activities and motivational interviewing (MI). The investigators will intervene at both the community and individual level. At the individual level, they will provide MICUNAY to adolescents. At the community level, they will provide discussion of AOD prevention at Community Wellness Gatherings (CWG). This work is important because they will gain an understanding of how well a tradition-based healing program that integrates MI works to prevent AOD use among urban AI/AN youth.

DETAILED DESCRIPTION:
American Indian/Alaska Native (AI/AN) youth report higher rates of alcohol and drug (AOD) use, greater frequency and intensity of AOD use, earlier first AOD use, and much higher alcohol-related mortality than other racial/ethnic groups in the U.S. Data regarding urban AIs/ANs are limited; however, one study found that at-risk AIs/AN adults in an urban setting report an earlier onset of alcohol, marijuana, methamphetamine, and other drug use compared to all other ethnic/racial groups within LA County. This proposal responds to PAR-11-346, Interventions for Health Promotion and Disease Prevention in Native American Populations, which is focused on developing, adapting, and testing the effectiveness of health promotion prevention interventions in Native American populations. The two co-PI's provide a unique blend of expertise that has resulted in the development of an innovative preliminary protocol for AI/AN youth: Motivational Interviewing and Culture for Urban Native American Youth (MICUNAY), which integrates traditional healing approaches with motivational interviewing (MI). Dickerson is an Alaska Native (Inupiaq) new investigator who worked with the AI/AN community to obtain community-based perspectives on decreasing AOD use and mental health problems. D'Amico is internationally recognized for her work focused on the development and testing of MI interventions targeting AOD use for culturally diverse adolescents across different settings. Dickerson and colleagues have demonstrated the need for culturally-appropriate interventions for AI/AN youth. His two community-based projects found that there is a lack of programs integrating tradition-based healing with evidenced based treatments (EBTs), and this was cited as a significant barrier to seeking care within urban AI/AN populations. Therefore, MICUNAY will integrate tradition-based healing with MI. It consists of 6 weekly 1-hour sessions (3 MI AOD sessions and 3 tradition activity sessions). This proposal also incorporates a multi-system intervention approach. At the individual level, the investigators will provide MICUNAY to urban AI/AN youth. At the community level, they will discuss AOD use and AOD prevention among AI/AN youth at existing Community Wellness Gatherings (CWG). The proposed 5-year study will consist of two main components: 1) A Developmental Phase in which they conduct focus groups across two clinical sites in Los Angeles and Oakland with the community to establish feasibility and sustainability of delivery, 2) A randomized controlled trial comparing youth who only attend a CWG (n=100) to youth who attend a CWG plus receive MICUNAY (n=100). The investigators will compare outcomes at 3- and 6-month follow-up to determine (a) whether clinically significant changes in AOD expectancies, perceived prevalence of peer AOD use, alcohol consumption, marijuana and other drug use, and related consequences occur; (b) whether clinically significant changes in physical, social, emotional, and functional well-being as well as spirituality and cultural identification occur, and (c) if reductions occur, estimate effect sizes for the CWG group and the CWG plus MICUNAY group. This study substantially extends work with AI/AN youth by intervening at both the community and individual level, and developing and testing an integrated tradition-based AOD MI group intervention for urban AI/AN youth.

ELIGIBILITY:
Inclusion Criteria:

* identify as Native American
* age 14-18

Exclusion Criteria:

* just need to meet inclusion criteria

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D'Amico, PhD, Principal Investigator — RAND; Daniel Dickerson, D.O., M.P.H, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - United American Indian Involvement, Inc, Los Angeles, California
  - American Indian Child Resource Center, Oakland, California

REFERENCES:
- [Background] D'Amico EJ, Tucker JS, Miles JN, Ewing BA, Shih RA, Pedersen ER. Alcohol and marijuana use trajectories in a diverse longitudinal sample of adolescents: examining use patterns from age 11 to 17 years. Addiction. 2016 Oct;111(10):1825-35. doi: 10.1111/add.13442. Epub 2016 Jun 14. PMID 27130360
- [Background] Ellickson PL, McCaffrey DF, Ghosh-Dastidar B, Longshore DL. New inroads in preventing adolescent drug use: results from a large-scale trial of project ALERT in middle schools. Am J Public Health. 2003 Nov;93(11):1830-6. doi: 10.2105/ajph.93.11.1830. PMID 14600049
- [Background] D'Amico EJ, Miles JN, Stern SA, Meredith LS. Brief motivational interviewing for teens at risk of substance use consequences: a randomized pilot study in a primary care clinic. J Subst Abuse Treat. 2008 Jul;35(1):53-61. doi: 10.1016/j.jsat.2007.08.008. Epub 2007 Nov 26. PMID 18037603
- [Background] Phinney, J. S., & Ong, A. D. (2007). Conceptualization and measurement of ethnic identity: Current status and future directions. Journal of Counseling Psychology, 54(3), 271.
- [Background] Ponterotto, J. G., Gretchen, D., Utsey, S. O., Stracuzzi, T., & Saya Jr, R. (2003). The multigroup ethnic identity measure (MEIM): Psychometric review and further validity testing. Educational and Psychological Measurement, 63(3), 502-515.
- [Background] Brown RA, Dickerson DL, D'Amico EJ. Cultural Identity Among Urban American Indian/Alaska Native Youth: Implications for Alcohol and Drug Use. Prev Sci. 2016 Oct;17(7):852-61. doi: 10.1007/s11121-016-0680-1. PMID 27450682
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Derived] Dickerson DL, Parker J, Johnson CL, Brown RA, D'Amico EJ. Recruitment and retention in randomized controlled trials with urban American Indian/Alaska Native adolescents: Challenges and lessons learned. Clin Trials. 2021 Feb;18(1):83-91. doi: 10.1177/1740774520971774. Epub 2020 Nov 24. PMID 33231130

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Given the importance to our partnering Native communities that every teen receive some culturally relevant intervention, our "control" group was not the standard control that is often seen in RCTs. Our control group comprised a large cultural event (Community Wellness Gathering or CWG) designed to connect adolescents with their heritage and AI/AN resources in their community. The intervention group received the CWG + MICUNAY.
Groups:
- Community Wellness Gathering + MICUNAY: Some participants randomized to MICUNAY, a three session workshop focused on discussions about how to make healthy choices using motivational interviewing, and providing a cultural activity.
  MICUNAY: MICUNAY is a three session workshop focused on discussions about how to make healthy choices using motivational interviewing, and providing a cultural activity.
Period: Overall Study
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Started | 70 | 115
Completed | 56 | 72
Not Completed | 14 | 43
Not completed — Lost to Follow-up | 14 | 43

BASELINE CHARACTERISTICS:
Population: Participants were aged 14-18 and self-identified as (or parents identified them as) American Indian/Alaska Native.
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY | Total
Number analyzed (Participants) | 70 | 115 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] — Asked how old they were.
  years | 15.51 (1.18) | 15.66 (1.41) | 15.61 (1.33)
Sex: Female, Male [Count of Participants; unit: Participants] — Asked participants their gender.
  Participants
    Female | 48 | 47 | 95
    Male | 22 | 68 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — We ask about a person's ethnicity to create statistics about ethnicity and to present other estimates by ethnic group.
  Participants
    Hispanic or Latino | 28 | 55 | 83
    Not Hispanic or Latino | 42 | 60 | 102
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — We ask about a person's race to create statistics about race and to present other estimates by race group.
  Participants
    American Indian or Alaska Native | 39 | 70 | 109
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 2 | 4 | 6
    White | 1 | 3 | 4
    More than one race | 21 | 22 | 43
    Unknown or Not Reported | 6 | 15 | 21
Minimum of Graduated from High School (mother) [Count of Participants; unit: Participants] — We asked study participants via baseline survey if mother was at least a high school graduate. Measure is an indicator of family socioeconomic status.
  Participants | 49 | 71 | 120
Minimum of Graduated from High School (father) [Count of Participants; unit: Participants] — We asked study participants via baseline survey if father was at least a high school graduate. Measure is an indicator of family socioeconomic status.
  Participants | 39 | 55 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used Alcohol From Baseline to 6 Months
Description: For this study, we created a dichotomous indicator of whether adolescents reported any use of alcohol. This is because alcohol use rates are typically lower in younger adolescents, leading to highly skewed distributions in continuous variables.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Count of Participants; unit: Participants
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
Participants | 22 | 33

2. Primary Outcome: Number of Participants Who Used Marijuana From Baseline to 6 Months
Description: For this study, we created a dichotomous indicator of whether adolescents reported any use of marijuana. This is because marijuana use rates are typically lower in younger adolescents, leading to highly skewed distributions in continuous variables.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Count of Participants; unit: Participants
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
Participants | 22 | 32

3. Secondary Outcome: Number of Participants Who Reported Consequences of Alcohol Use
Description: Adolescents reported on the alcohol consequences they had experienced in past three months. Consequences are based on DSM-IV criteria with 7 items for alcohol (e.g., missed school or work). For this analysis we created dichotomous indicators of whether adolescents reported any consequences from alcohol.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Count of Participants; unit: Participants
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
Participants | 23 | 37

4. Secondary Outcome: Number of Participants Who Reported Consequences of Marijuana Use
Description: Adolescents reported on the marijuana consequences they had experienced in past three months. Consequences are based on DSM-IV criteria with 5 items for marijuana (e.g., had difficulty concentrating). For this analysis we created dichotomous indicators of whether adolescents reported any consequences from marijuana.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Count of Participants; unit: Participants
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
Participants | 23 | 35

5. Secondary Outcome: Change in Intentions to Use - Alcohol
Description: Three separate items assessed whether adolescents believed they would drink any alcohol, use any marijuana, or smoke a cigarette in the next six months (1="definitely yes" to 4="definitely no").
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 1.84 (1.04) | 1.65 (0.96)

6. Secondary Outcome: Change in Intentions to Use - Cigarettes
Description: as for outcome 5
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 1.77 (1.23) | 1.66 (1.14)

7. Secondary Outcome: Change in Intentions to Use - Marijuana
Description: as for outcome 5
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 2.03 (1.14) | 1.92 (1.15)

8. Secondary Outcome: Change in Alcohol Resistance Self-efficacy
Description: Alcohol resistance self-efficacy (RSE) for alcohol was defined as the average of four items rated from "I would definitely use" to "I would definitely not use" based on different situations (e.g., if my best friend were using; you were bored at party; your friend gives you a drink). RSE ranged from 1 to 4; higher scores indicated greater RSE.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 3.00 (1.06) | 2.95 (1.09)

9. Secondary Outcome: Change in Peer Influence - Alcohol
Description: Three separate items assessed how often adolescents spend time around teens who drink, use marijuana, or smoke cigarettes (1 = "never" to 4 = "often").
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 1.76 (0.94) | 1.76 (0.99)

10. Secondary Outcome: Change in Peer Influence - Marijuana
Description: as for outcome 9
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 2.14 (1.18) | 2.04 (1.18)

11. Secondary Outcome: Change in Peer Influence - Cigarettes
Description: as for outcome 9
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 1.53 (0.93) | 1.54 (0.83)

12. Secondary Outcome: Change in Intentions to Participate in Traditional Practices
Description: Adolescents reported how likely they were to participate in >20 different traditional practices (e.g., going to Pow Wows, prayer, playing Native hand or stick games) in the next six months (1="definitely yes" to 4="definitely no").
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 2.71 (0.96) | 2.68 (0.89)

13. Secondary Outcome: Change in Cultural Identification
Description: We assessed adolescents' AI/AN cultural pride and sense of belonging with the Multigroup Ethnic Identity Measure (MEIM), which has twelve items. Respondents are asked the degree to which they agree with statements such as, "I have a clear sense of my ethnic background and what it means to me" on a scale from 1 = "strongly disagree" to 5 = "strongly agree". Given that our prior focus group work indicated that many adolescents were of mixed ethnicity, and our focus was on AI/AN identity, we modified these items to focus on AI/AN heritage (e.g., "I have clear sense of my AI/AN identity and what it means to me").
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 3.11 (1.13) | 3.39 (1.14)

14. Secondary Outcome: Change in Spirituality/Happiness
Description: Spirituality and happiness were measured using a subset of ten items from the 12-item Functional Assessment of Chronic Illness Therapy-Fatigue-Spiritual Questions instrument, or FACIT-SP 12. Adolescents reported agreement with statements such as "I find comfort in my faith or spiritual beliefs" and "I feel a sense of harmony within myself." Two items that referred specifically to chronic illness were removed from the scale as they were not relevant for this study. Response options, which ranged from 1="not at all" to 5="very much," were averaged, with negative statements reversed such that higher scores indicated greater spirituality and happiness.
Time Frame: change from baseline to 6 months
Population: American Indian/Alaska Native adolescents aged 14-18.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
Number analyzed (Participants) | 70 | 115
score on a scale | 3.12 (1.24) | 3.29 (1.29)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Total Number of Participants at Risk was 185.
Arm/Group | Community Wellness Gatherings | Community Wellness Gathering + MICUNAY
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/115
Other Adverse Events (participants affected / at risk) | 0/70 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02290938/Prot_SAP_000.pdf
  • Informed Consent Form (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02290938/ICF_001.pdf